CLINICAL TRIAL: NCT01072487
Title: Capnography as an Adjunct to Standard Monitoring During Midazolam and Propofol Sedation for Colonoscopy
Brief Title: Capnography During Colonoscopy
Acronym: ColoCap
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Stefan von Delius, II. Medizinische Klinik der Technischen Universität München
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2681/10
Record Dates: First submitted 2010-02-17; First posted 2010-02-22 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Hypoxemia; Complications
Keywords: Safety; Sedation; Gastrointestinal endoscopy; Colonoscopy
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capnography (Experimental): Arm with capnographic monitoring
  Interventions: Procedure: Capnography
- Standard (No Intervention): Standard monitoring.

INTERVENTIONS:
Procedure: Capnography — Monitoring of the capnography curve for early detection of apnea
  Arms: Capnography

SUMMARY:
In the study the value of capnography for avoiding complications during sedation for colonoscopy is evaluated.

DETAILED DESCRIPTION:
In this randomized controlled trial the utility of capnography gets evaluated. Hypoxemia may occur during sedation with midazolam and propofol. Whether hypoxemia may be prevented by an additional capnographic monitoring is subject of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18
* Scheduled for colonoscopy with midazolam and propofol sedation

Exclusion Criteria:

* No informed consent
* ASA IV or V
* Pregnancy
* Prexisting hypotension, bradycardia or hypoxemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | From the start to the end of colonoscopy, i.e. from 0 h to approximately 2 h

SECONDARY OUTCOMES:
Further complications | From the start to the end of colonoscopy, i.e. from 0 h to approximately 2 h

CONTACTS AND LOCATIONS:
Overall Officials: Stefan von Delius, MD, Principal Investigator — Technical University of Munich
Locations (3):
- Germany (3):
  - Technische Universität München, Munich, Bavaria
  - Knappschaftskrankenhaus der Ruhr-Universität Bochum, Bochum
  - Deutsche Klinik für Diagnostik, Wiesbaden

REFERENCES:
- [Background] Qadeer MA, Vargo JJ, Dumot JA, Lopez R, Trolli PA, Stevens T, Parsi MA, Sanaka MR, Zuccaro G. Capnographic monitoring of respiratory activity improves safety of sedation for endoscopic cholangiopancreatography and ultrasonography. Gastroenterology. 2009 May;136(5):1568-76; quiz 1819-20. doi: 10.1053/j.gastro.2009.02.004. PMID 19422079
- See also: II. Medizinische Klinik der Technischen Universität München — http://www.med2.med.tu-muenchen.de/